CLINICAL TRIAL: NCT04086823
Title: A Single Blind, Randomized, Placebo-controlled, Phase 2a, 2-cohort Study for the Evaluation of Safety and Efficacy of RZL-012 for Submental Fat Reduction in Healthy Volunteers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Raziel Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RZL-012-SMF-P2aUS-001
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2019-09

CONDITIONS: Submental Fat
MeSH Terms: interventions — RZL-012

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RZL-012 (Active Comparator): A single-treatment injection, multiple subcutaneous injections of RZL-012 administered into 48 sites in the submental fat (0.05/0.1mL per site):
  1. Up to 120mg administered at 48 sites in a volume of 0.05 ml at each injection site (total injected volume 2.4mL)
  2. Up to 240 mg administered at 48 sites in a volume of 1 ml at each injection site (total volume injected 4.8mL)
  Interventions: Drug: RZL-012
- Vehicle (Placebo Comparator): Subject receive a single-treatment injection. Multiple injections of the Placebo are administered at 48 sites (0.05/0.1mL per site) into the submental fat.
  Up to a total of 2.4 mL will be injected for placebo subjects enrolled during cohort 1.
  Up to a total of 4.8 mL will be injected for placebo subjects enrolled during cohort 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RZL-012 — Subcutaneous injection to the submental fat area
  Arms: RZL-012
Drug: Placebo — Placebo
  Arms: Vehicle

SUMMARY:
Twenty-Eight (28) subjects (12 for cohort 1 and 16 for cohort 2 ) will be included in the study. Subjects in each cohort will be injected with a different dose of RZL-012. The total of 28 subjects will be enrolled in 2 clinical sites.

DETAILED DESCRIPTION:
This is a single blinded, randomized, placebo-controlled, 2-cohort clinical study in healthy volunteers. Cohort 1 will be comprised of 8 active (RZL-012) and 4 placebo subjects. Cohort 2 will be comprised of 16 subjects wuth at least 4 placebo subjects. All subjects will receive a single dose of RZL-012 or vehicle into the submental area, after which they will be monitored for safety and efficacy during 84 days of follow-up.

Subjects will be blinded to study treatment while physicians will not be blinded.

The study will be composed of 2 treatment cohorts, 12 in cohort 1 and 16 in cohort 2.

The study will be conducted in 2 clinical sites. Per each study cohort, subjects will be randomized to receive active or placebo treatment according to a randomization program that will be prepared prior to study initiation. Each clinical site will have at least one active and one placebo treatment subject per each study cohorts. In case of slow enrollment in one of the sites, other sites may complete the enrollment of subjects in each cohort.

Cohort 1 (N=12) - Each subject will be dosed with up to 120 mg RZL-012 (depending on submental fat area) or vehicle.

Cohort 2 (N=16) - Each subject will be dosed with up to 240 mg RZL-012 (depending on submental fat area) or vehicle.

Treatment of cohort 2 will start following cohort 1 day 28 data. An independent Data Safety Monitoring Board (DSMB) will review safety and tolerability data for cohort 1 subjects, 28 days after injection, and decide whether it is safe to increase the dose for the next study cohort. The decision to proceed to the cohort 2 will be made within 30 days (28 days + 2 days) after injection of the last dosed subject in cohort 1.

The DSMB will be comprised of two independent MDs with expertise in the aesthetic area and in conduction of clinical trials.

In case of serious safety concerns (e.g. prolonged severe swelling or severe pain following injection) among cohort 1 subjects receiving the 120mg dose, sponsor and DSMB may decide to reduce or stay with the 120mg/subject dose level for cohort 2 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-65 years old.
2. Subjects with Body Mass Index <35
3. Subjects must have submental skin fold thickness greater than 1.5 cm as measured with calipers.
4. Males must be willing to be clean shaved for all study visits.
5. Patient weight must be stable (no fluctuation of >15 pounds in the past year)
6. Males or females in the age of fertility agree to use a double-barrier contraceptive device (e.g., condom and spermicide) for 4 weeks after treatment with RZL 012.
7. Subjects must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
8. Subjects must sign an IRB approved informed consent indicating they are aware of the investigational nature of the study.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from study participation:

1. Unable to tolerate subcutaneous injection.
2. Pregnant or lactating women.
3. Subjects with dysfunctional gallbladder activity, e.g. underwent cholecystectomy or cholecystitis.
4. Any uncontrolled systemic disease -a potential patient in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study
5. Treatment with botulinum toxin injections in the neck or chin area within 6 months before screening.
6. Excessive submental skin laxity.
7. Any Scars, unshaven hair, tattoos or jewelry on or near the proposed treatment area
8. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study
9. An active dermatitis or open wound in the proposed treatment area
10. An active bacterial, fungal, or viral infection in the proposed treatment area
11. Pre-existing skin condition in the submental region that may confound evaluation or analysis, at investigator discretion
12. Previously treated with focused ultrasound, radiofrequency, cryolipolysis, liposuction, sodium deoxycholate to the submental region within the previous 6 months
13. Pre-existing neurological or gastrointestinal condition leading to dysphagia, dysphonia or facial nerve palsy
14. Pre-existing medical condition other than increased submental fat that may result in increased submental fullness such as but not limited to thyroid enlargement, goiter, cervical lymphadenopathy etc., at investigator discretion
15. Must not have a planned fat reduction procedure of any variety to the submental region for the duration of the study
16. Must not have planned significant alterations in diet or physical activity that may result in significant fluctuations in weight.
17. Subjects with medication or history of coagulopathy.
18. Allergic subjects to Bendaryl.
19. Subjects treated chronically at least 3 months prior to study entry with systemic steroids or immunosuppressive drugs.
20. Subjects treated chronically at least one week prior to study entry with Non-Steroidal Anti-Inflammatory Drugs (NSAIDs).
21. Current participation or participation within 3 months prior to the start of this study in a drug or other investigational research study.
22. Claustrophobia or MRI incompatible device or implant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- DeNova Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The safety and efficacy of exposed subjects to RZL-012 were compared to exposed subjects with placebo
Groups:
- RZL-012 Cohort 1: A single-treatment injection, multiple subcutaneous injections of RZL-012 administered into 48 sites in the submental fat (0.05mL per site):
  1. Up to 120mg administered at 48 sites in a volume of 0.05 ml at each injection site (total injected volume 2.4mL)
- Vehicle Cohort 1: Subject receive a single-treatment injection. Multiple injections of the Placebo are administered at 48 sites (0.05mL per site) into the submental fat.
  Up to a total of 2.4 mL will be injected for placebo subjects enrolled during cohort 1.
  Placebo: Placebo
- RZL-012 Cohort 2: A single-treatment injection, multiple subcutaneous injections of RZL-012 administered into 48 sites in the submental fat (0.1mL per site):
  Up to 240 mg administered at 48 sites in a volume of 1 ml at each injection site (total volume injected 4.8mL)
  RZL-012: Subcutaneous injection to the submental fat area
- Vehicle Cohort 2: Subject receive a single-treatment injection. Multiple injections of the Placebo are administered at 48 sites (0.1mL per site) into the submental fat.
  Up to a total of 4.8 mL will be injected for placebo subjects enrolled during cohort 2.
Period: Overall Study
Arm/Group | RZL-012 Cohort 1 | Vehicle Cohort 1 | RZL-012 Cohort 2 | Vehicle Cohort 2
Started | 8 | 4 | 10 | 6
Completed | 8 | 4 | 10 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline is defined as the last available and evaluable parameter value before and closest to the injection.
Groups:
- RZL-012 Cohort 1: A single-treatment injection, multiple subcutaneous injections of RZL-012 administered into 48 sites in the submental fat (0.05mL per site):
  Up to 120mg administered at 48 sites in a volume of 0.05 ml at each injection site (total injected volume 2.4mL)
  RZL-012: Subcutaneous injection to the submental fat area
- Vehicle Cohort 1: Subject receive a single-treatment injection. Multiple injections of the Placebo are administered at 48 sites (0.05mL per site) into the submental fat.
  Up to a total .of 2.4 mL will be injected for placebo subjects enrolled during cohort 2.
  Placebo: Placebo
- Vehicle Cohort 2: Subject receive a single-treatment injection. Multiple injections of the Placebo are administered at 48 sites (0.1mL per site) into the submental fat.
  Up to a total of 4.8 mL will be injected for placebo subjects enrolled during cohort 2.
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | RZL-012 Cohort 1 | Vehicle Cohort 1 | RZL-012 Cohort 2 | Vehicle Cohort 2 | Total
Number analyzed (Participants) | 8 | 4 | 10 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (6.8) | 57.5 (8.2) | 43.3 (9.5) | 48.8 (10.2) | 49.65 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9 | 6 | 24
  Male | 2 | 1 | 1 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 4 | 9 | 5 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 8 | 4 | 9 | 6 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 4 | 10 | 6 | 28

OUTCOME MEASURES:

1. Primary Outcome: Safety: Adverse Events Follow up
Description: To evaluate the safety of RZL-012 subcutaneous injections in the submental area, relative to placebo, as assessed by spontaneous adverse event reports and post injection evaluation of subjects. Specifically, Pain, Induration, Bruising, Erythema and Edema will be closely followed up following treatment.
Time Frame: 0-84 days
Population: Safety Analysis consist of all enrolled subjects who received the study treatment, (exposed population), vs. placebo treated subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Vehicle: Subject receive a single-treatment injection. Multiple injections of the Placebo are administered at 48 sites (0.05mL per site) into the submental fat.
  Up to a total of 2.4 mL will be injected for placebo subjects enrolled during cohort 1.
  Placebo: Placebo
- RZL-012 Cohort 2: A single-treatment injection, multiple subcutaneous injections of RZL-012 administered into 48 sites in the submental fat (0.1mL per site):
  Up to 240 mg administered at 48 sites in a volume of 1 ml at each injection site (total volume injected 4.8mL)
Arm/Group | RZL-012 Cohort 1 | Vehicle | RZL-012 Cohort 2 | Vehicle Cohort 2
Number analyzed (Participants) | 8 | 4 | 10 | 6
Participants | 8 | 4 | 10 | 6

2. Secondary Outcome: Physician's Global Assessment
Description: Evaluation of treatment efficacy by using Physician's global assessment questionnaire for active vs. placebo subjects, on study Day 84
Time Frame: 0-84 days
Population: Subjects were analysed according to the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | RZL-012 Cohort 1 | Vehicle Cohort 1 | RZL-012 Cohort 2 | Vehicle Cohort 2
Number analyzed (Participants) | 8 | 4 | 10 | 6
Participants
  Subjects experienced improvement (Score =0 (completely clear) , 1, 2, 3, Score=4(slight improvement) | 7 | 0 | 10 | 0
  Subjects that experienced no improvement = Score 5 (no Change) | 1 | 4 | 0 | 6

3. Secondary Outcome: Efficacy: MRI Volume Reduction
Description: Reduction from baseline in submental fat volume, as measured with MRI, in RZL-012 treated subjects vs. placebo treated subjects on Day 84 following injection.
Time Frame: 0-84 days
Population: The efficacy in the MRI was divided to per treated doses cohorts
Measure: Mean (Standard Deviation); unit: percentage of volume reduction high dose
Groups:
- RZL-012: A single-treatment injection, multiple subcutaneous injections of RZL-012 administered into 48 sites in the submental fat (0.05/0.1mL per site):
  1. Up to 120mg administered at 48 sites in a volume of 0.05 ml at each injection site (total injected volume 2.4mL)
  2. Up to 240 mg administered at 48 sites in a volume of 1 ml at each injection site (total volume injected 4.8mL)
  RZL-012: Subcutaneous injection to the submental fat area
- Vehicle: Subject receive a single-treatment injection. Multiple injections of the Placebo are administered at 48 sites (0.05/0.1mL per site) into the submental fat.
  Up to a total of 2.4 mL will be injected for placebo subjects enrolled during cohort 1.
  Up to a total of 4.8 mL will be injected for placebo subjects enrolled during cohort 2.
  Placebo: Placebo
Arm/Group | RZL-012 | Vehicle
Number analyzed (Participants) | 18 | 10
percentage of volume reduction high dose
  Cohort 2 High Dose (BioClinica Analysis): number analyzed (Participants) | 10 | 6
  Cohort 2 High Dose (BioClinica Analysis) | -12.5 (8) | 0.7 (8.5)
  Cohort 1 Low Dose (Bioclinica Analysis): number analyzed (Participants) | 8 | 4
  Cohort 1 Low Dose (Bioclinica Analysis) | -6.4 (11) | -5.7 (3)

4. Secondary Outcome: Efficacy: Improvement in Face Satisfaction Questionnaire - A Score From 0 (Worst) to 100 (Best) Marks the Subject's Satisfaction
Description: Improvement from baseline in the Faceq satisfaction questionnaire rating score in RZL-012 treated subjects vs. placebo treated subjects on day 84.
Time Frame: 0-84 days
Population: The questionnaire efficacy included all exposed population to RZL-012 vs. all treated subjects by placebo
Measure: Mean (Standard Deviation); unit: change in scores on a scale
Arm/Group | RZL-012 Cohort 1 | Vehicle Cohort 1 | RZL-012 Cohort 2 | Vehicle Cohort 2
Number analyzed (Participants) | 8 | 4 | 10 | 6
change in scores on a scale | 34.8 (10) | -3.8 (29.2) | 38.5 (25) | -1.2 (16.3)

ADVERSE EVENTS:
Time Frame: 84 days
Description: All reported adverse events were related to injection site condition.
Arm/Group | RZL-012 Cohort 1 | Vehicle Cohort 1 | RZL-012 Cohort 2 | Vehicle Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 4/4 | 10/10 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RZL-012 Cohort 1 (N=8) | Vehicle Cohort 1 (N=4) | RZL-012 Cohort 2 (N=10) | Vehicle Cohort 2 (N=6)
Edema (General disorders) | 4 | 2 | 6 | 3 — General disorders and administration site condition
Induration (General disorders) | 4 | 2 | 6 | 3 — General disorders and administration site condition
Injection site bruising (General disorders) | 5 | 3 | 7 | 3 — General disorders and administration site condition
Injection site erythema (General disorders) | 4 | 2 | 3 | 1 — General disorders and administration site condition
Injection site edema (General disorders) | 0 | 0 | 1 | 0 — General disorders and administration site condition
Injection site pain (General disorders) | 4 | 2 | 4 | 2 — General disorders and administration site condition
Bruising sensation (Nervous system disorders) | 2 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT04086823/Prot_SAP_000.pdf